CLINICAL TRIAL: NCT00290654
Title: Twin Cities Brachytherapy Study for Ductal Carcinoma in Situ A Phase II Trial
Brief Title: Internal Radiation Therapy After Lumpectomy in Treating Women With Ductal Carcinoma in Situ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit further patients.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002LS097; UMN-0211M35761 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Tamoxifen; Mastectomy, Segmental; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lumpectomy with Brachytherapy (Experimental): Patients with ductal carcinoma in situ (DCIS, a non-invasive form of breast cancer) treated with standard lumpectomy/brachytherapy following by radiation using the MammoSite (FDA approved a balloon-catheter device placed in the lumpectomy cavity through which high dose radiation is delivered). Tamoxifen may be used postoperatively at the discretion of the treating physicians and patient.
  Interventions: Drug: Tamoxifen; Procedure: Lumpectomy; Radiation: brachytherapy

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen may be used postoperatively at the discretion of the treating physicians and patient
Procedure: Lumpectomy — A standard lumpectomy will be performed with an attempt to remove at least 1 cm of gross margin around the DCIS.
Radiation: brachytherapy — Treatment will be given in 10 fractions of 3.4 Gy per fraction twice a day, with a minimum of 6 hours between fractions. In general, brachytherapy will start between 2 - 5 days of implant. All treatments will be done using a commercially available HDR and 192Ir radioactive sources.

SUMMARY:
RATIONALE: Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving internal radiation therapy using a special radiation therapy device may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well internal radiation therapy after lumpectomy works in treating women with ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the ipsilateral breast tumor recurrence rate in women with ductal carcinoma in situ undergoing lumpectomy followed by brachytherapy using the MammoSite^® Radiation Therapy System.

Secondary

* Determine the early and late complication rates and cosmetic outcome in these patients after treatment.

OUTLINE: Patients undergo lumpectomy. Patients with negative tumor margins* (no ink on tumor) undergo placement of the MammoSite^® Radiation Therapy System at the time of lumpectomy or within 4 weeks after surgery.

NOTE: *If positive margins are present, the surgeon may elect to resect the positive margins and then insert a new MammoSite® device if all other eligibility criteria are met.

Beginning 2-5 days after placement of the MammoSite^®, patients undergo brachytherapy through the MammoSite^® twice daily for 5 days (a total of 10 fractions).

After completion of study treatment, patients are followed periodically for ≥ 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Ductal carcinoma in situ (DCIS) confirmed by excisional or needle biopsy
* Size: < 3 cm on mammogram
* Unicentric disease
* Ability to place MammoSite device at time of lumpectomy or within 4 weeks of lumpectomy
* Patient Age: ≥ 18 years, no upper limit
* Life expectancy > 5 years

Exclusion Criteria:

* Prior history of cancer other than basal or squamous cell skin cancer or in situ cancer of the cervix
* Pregnant or breast feeding
* Multicentric disease
* Diagnosis of collagen vascular diseases, such as systemic lupus erythematosis, scleroderma, or dermatomyositis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Tuttle, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients wereinvited to participate in the study by their physician, who explained the details of the trial and obtained informed consent. Patients who met the eligibility criteria and signed the appropriate consent were entered into the study before the MammoSite device was inserted.
Pre-assignment Details: A total of 45 subjects were enrolled. Four subjects did not receive accelerated partial breast irradiation because the minimum distance from the skin to the internal radiation device was <5mm and is associated with poor cosmetic results.
Groups:
- MammoSite Treatment Group: Patients with ductal carcinoma in situ (DCIS, a non-invasive form of breast cancer) treated with standard lumpectomy/brachytherapy following by radiation using the MammoSite (FDA approved a balloon-catheter device placed in the lumpectomy cavity through which high dose radiation is delivered). Tamoxifen may be used postoperatively at the discretion of the treating physicians and patient.
Period: Overall Study
Arm/Group | MammoSite Treatment Group
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MammoSite Treatment Group
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 54 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Ipsilateral Breast Tumor Recurrence
Description: Count of patients with early stage breast cancer who developed an ipsilateral breast tumor recurrence (IBTR) and failed after receiving breast-conserving therapy.
Time Frame: 1 year after treatment
Measure: Number; unit: participants
Groups:
- Evaluable Patients: Number of patients who had lumpectomy and completed partial breast radiation using a unique balloon-catheter application device.
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 41
participants | 0

2. Primary Outcome: Number of Patients With Ipsilateral Breast Tumor Recurrence
Description: as for outcome 1
Time Frame: 5 years after treatment
Measure: Number; unit: participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 41
participants | 4

3. Secondary Outcome: Percentage of Patients Who Experienced Complications
Description: Complications to be measured include: breast tenderness/pain,reddening of the skin, bruising, formation of blood or fluid under the skin, skin ulceration, infection, discoloration of the skin, development of telangiectasia (spider veins), hardening of the breast tissue, and retraction of the breast tissue.
Time Frame: within 6 months of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 41
percentage of participants | 65.8

4. Secondary Outcome: Percentage of Patients Who Experienced Complications
Description: as for outcome 3
Time Frame: more than 6 months after treatment, for up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 41
percentage of participants | 24.4

5. Secondary Outcome: Percentage of Physicians Judging the Cosmetic Outcome as Good or Excellent
Description: The following items will be evaluated by comparing the treated breast with the untreated breast: overall cosmetic result; appearance of the surgical scar; breast size; breast shape; nipple position; and shape of areola. In scoring these items, a 4-point scale will be used, classifying the results into one of the following categories: "0" representing an excellent result; "1" a good result; "2" a fair result; and "3" a poor result.
Time Frame: 6 months after treatment
Measure: Number; unit: percentage of physicians
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 41
percentage of physicians | 100

6. Secondary Outcome: Percentage of Physicians Judging the Cosmetic Outcome as Good or Excellent
Description: as for outcome 5
Time Frame: 12 months after treatment
Measure: Number; unit: percentage of physicians
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 41
percentage of physicians | 86.7

7. Secondary Outcome: Percentage of Patients Judging the Cosmetic Outcome as Good or Excellent
Description: as for outcome 5
Time Frame: 6 months after treatment
Measure: Number; unit: percentage of participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 41
percentage of participants | 96.8

8. Secondary Outcome: Percentage of Patients Judging the Cosmetic Outcome as Good or Excellent
Description: as for outcome 5
Time Frame: 12 months after treatment
Measure: Number; unit: percentage of participants
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 41
percentage of participants | 92.3

ADVERSE EVENTS:
Arm/Group | MammoSite Treatment Group
Serious Adverse Events (participants affected / at risk) | 1/41
Other Adverse Events (participants affected / at risk) | 28/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MammoSite Treatment Group (N=41)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MammoSite Treatment Group (N=41)
Breast tenderness/pain - early onset (Injury, poisoning and procedural complications) | 11
Breast tenderness/pain - late onset (Injury, poisoning and procedural complications) | 4
Erythema - early onset (Injury, poisoning and procedural complications) | 11
Hematoma/seroma - early onset (Injury, poisoning and procedural complications) | 5
Infection - early onset (Infections and infestations) | 4
Pigmentation - early onset (Skin and subcutaneous tissue disorders) | 8
Telangiectasia - late onset (Skin and subcutaneous tissue disorders) | 4
Induration - early onset (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes